CLINICAL TRIAL: NCT04021329
Title: Efficacy of Eye Movement Desensitization & Reprocessing Versus Cognitive Behavioral Therapy in Post-Traumatic Stress and Depressive Disorders: Study Protocol for a Randomized Controlled Trial
Brief Title: Efficacy of Eye Movement Desensitization & Reprocessing Versus Cognitive Behavioral Therapy in Post-Traumatic Stress and Depressive Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khushal Khan Khattak Univeristy, Karak, Pakistan (Other)
Responsible Party: Principal Investigator, Dr. Anwar Khan, Assistant Professor, Khushal Khan Khattak Univeristy, Karak, Pakistan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KhushalKhanKhattakU
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Efficacy of Psychotherapy
Keywords: Post-traumatic Stress Disorder, Major Depressive Disorder, Comorbidity, Eye Movement Desensitization & Reprocessing, Cognitive Behavioral Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: The current study will be a two arms cross over Randomized Controlled Trial (RCT) with Repeated Measures.
  Moreover, the Consolidated Standards of Reporting Trials (CONSORT) group flow diagram and SPIRIT Checklist will be followed to carry out and report this study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR Therapy (Other): One arm will be a group subjected to EMDR Therapy
  Interventions: Behavioral: CBT Therapy
- CBT Therapy (Other): other arm will be a group subjected to CBT Therapy
  Interventions: Behavioral: CBT Therapy

INTERVENTIONS:
Behavioral: CBT Therapy — information added previously
  Other Names: EMDR Therapy

SUMMARY:
Post-Traumatic Stress Disorder(PTSD) develops after exposure to or witnessing traumatic events. PTSD is highly comorbid and individuals with PTSD usually report Major Depressive Disorder(MDD). Common treatment choices for PTSD and MDD are either EMDR or CBT, however, little is known about their comparative efficacy, especially in Pakistan. Therefore, this Randomized Controlled Trial(RCT) aims at determining the comparative efficacy of EMDR vs CBT in Pakistan. This study will also examine the association between reduction in symptoms of PTSD and MDD over course of treatment. In this regard, two arms Crossover Randomized Controlled Trial(RCT) with Repeated Measures Design will be selected. This study will be conducted at two rehabilitation centres and patients will be screened at Time:01, baseline; Time:02, during treatment; Time:03, post treatment and Time:04, 06 months follow-up. All analyses will be performed according to intention-to-treat principle. Variations in symptoms will be analysed by using descriptive statistics, χ2 tests, t-tests, and one way ANOVA. To examine changes in PTSD and MDD across time and to check efficacy of each treatment, a series of Linear Mixed Models will be run. Furthermore, a series of multi-level lagged mediation analysis will be performed to check bi-directional mediation between changes PTSD and MDD over time. This protocol has outlined the rationale for determining efficacy of EMDR and CBT in Pakistan. It will help in answering a broad range of questions concerning efficacy of newly developed evidence-based treatments. Moreover, it may also guide future research on the treatment of PTSD and MDD in the developing countries.

DETAILED DESCRIPTION:
Study Background: Post-Traumatic Stress Disorder (PTSD) and its associated comorbidities develop after exposure to the traumatic events. In the recent years a global increase in the rate of PTSD and its comorbidities has been observed, especially in the developing countries like Pakistan that is continually suffering from war on terrorism, domestic violence, coupled by poverty and cultural constraints. Due to increasing rates of PTSD and lack of treatment facilities in Pakistan, it is imperative to find a mechanism for controlling mental illnesses in Pakistan. This situation also motivates research on testing the efficacy of modern psychotherapies like EMDR and CBT. Aim: The present study aims at determining the efficacy of EMDR by comparing it with CBT for the treatment of PTSD and comorbid Major Depressive Disorder(MDD) in Pakistan. Research Design: A two arms Crossover Randomized Controlled Trial (RCT) with Repeated Measures Design will be selected. Consolidated Standards of Reporting Trials (CONSORT) group flow diagram will be followed to carry out and report this study. Participants and Setting: This study will be conducted at two rehabilitation centres situated in the district Peshawar, Pakistan. A formal sample size cannot be calculated at this stage because the exact number of PTSD patients located in the selected area is not known. However, participants will be recruited through consecutive sampling technique with a rolling recruitment strategy. The outdoor and indoor patients, who pass exclusion criteria and are positively screen for PTSD symptoms will be recruited for this study. The sample size will be 100 patients depending on the availability and willingness of patients. The patients will be randomly allocated either to EMDR or CBT with an allocation ratio of 1:1. Interventions: Patients will be screened (Time: 01, baseline) then they will undertake 06 psychotherapy sessions. After completing 06 sessions, patients will be assessed (Time: 02, during treatment). Additional 08 psychotherapy sessions will be carried out and after completing 14 sessions, the patients will be once again assessed (Time: 03, post treatment) and then assessed after 06 months (Time: 04, follow-up). Statistical Analyses: All analyses will be performed according to the intention-to-treat (ITT) principle. Variations in symptoms with regard to demographic/baseline characteristics will be analysed by using descriptive statistics, χ2 tests for categorical variables, t-tests, and one way ANOVA for continuous variables. Non-inferiority testing will be used to know whether EMDR is not worse than CBT. To examine changes in PTSD and its associated comorbidities across Time :01, Time: 02, Time: 03 and Time :04 and to check the efficacy of each treatment, a series of Linear Mixed Models, with Maximum Like hood Estimation will be run, including main effects of treatment and time and the interaction effects of treatment*time. Moreover, a series of multi-level lagged mediation analysis along with moderated mediation analysis will be performed to check the bi-directional mediation between changes PTSD (as mediator) and changes in outcome variables (comorbid symptoms) over time. Means and standard deviations will be used to compute effect sizes (Cohen's d) for pre and post treatment and 6 months follow up

ELIGIBILITY:
Exclusion Criteria:

The following patients will be excluded:

1. Patients below the age of 18 years and above 60 years as this study is not on children or older patients;
2. Patients who can't move their hands and eyes/or can't perform basic movements;
3. Patients who are unconscious for longer periods and unable to recover consciousness;
4. Patients not meeting the basic screening criteria of PTSD/ PTSD is not the main problem;
5. Patients with severe intellectual impairments, since such patients are difficult to communicate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Measurement of Change in the symptoms of Post Traumatic Stress Disorder | 1st week (Baseline/pre-treatment screening, T-1); six weeks (during treatment screening, T-2); 12 weeks (post-treatment assessment, T-3). Finally, three months (follow up assessment, T-4).
  Clinician-Administered Post Traumatic Stress Disorder Scale-5 (Weathers, Blake, et al., 2013) These diagnostic tools will be used to assess the symptoms of Post Traumatic Stress Disorder. Any changes in the level of PTSD will be noted with respect to Pre, Mid and Post treatment stages The total symptom severity score is calculated by summing severity scores for the 20
  * Criterion A (items 1-5); (Exposure to actual or threatened death)
  * Criterion B (items 6-7); (Presence of intrusion symptoms associated with the traumatic events)
  * Criterion C (items 8-14); (Persistent avoidance of stimuli associated with the traumatic events)
  * Criterion D (items 15-20). (Negative alterations in cognitions and mood associated with the traumatic events) Severity Rating 0. Absent:
    1. Mild / subthreshold:.
    2. Moderate / threshold:
    3. Severe / markedly elevated:
    4. Extreme / incapacitating:
Measurement of Socio Demographic Profile | 1st week at start of treatment, i.e, from date of randomization
  Socio-demographic characteristics of the patients, like age, gender, marital status, occupation and social background

SECONDARY OUTCOMES:
Measurement of Change in the symptoms of major depression | 1st week (Baseline/pre-treatment screening, T-1); six weeks (during treatment screening, T-2); 12 weeks (post-treatment assessment, T-3). Finally, three months (follow up assessment, T-4).
  Beck Depression Inventory-II (Steer, Ball, Ranieri, & Beck, 1999; Beck, Ward, Mendelson, Mock, & Erbaugh, 1961) This Inventory will be used to assess the symptoms of Major Depressive Disorder. Any changes in the level of Major Depression will be noted with respect to Pre, Mid and Post treatment stages Each of the 21 items corresponding to a symptom of depression is summed to give a single score for the Beck Depression Inventory-II. There is a four-point scale for each item ranging from 0 to 3. On two items (16 and 18) there are seven options to indicate either an increase or decrease of appetite and sleep. Cut-off score guidelines for the BDI-II are given with the recommendation that thresholds be adjusted based on the characteristics of the sample, and the purpose for use of the Beck Depression Inventory-II. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe

CONTACTS AND LOCATIONS:
Locations (1):
- Anwar Khan, Karak, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
the data obtained will be published in peer reviewed journals
Supporting Information: Study Protocol, CSR
Time Frame: it will available next year on line
Access Criteria: will be on-line accessible